CLINICAL TRIAL: NCT05545930
Title: Analysis of Red Blood Cell Integrity and Efficiency of Recovery Using a Novel Surgical Sponge-Blood Recovery Device (ProCell)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: ProCell Surgical Inc. (Unknown)
Responsible Party: Principal Investigator, Mohammad El Diasty, Division Chief, Cardiac Surgery, UH Cleveland Medical Center, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY20220888
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Blood Recovery
Keywords: Open Heart Surgery; Heart Transplant; Lung Transplant; ProCell

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be blinded to the order of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hand Wrung (Active Comparator): Hand wrung refers to manually wringing surgical sponges by hand.
  Interventions: Procedure: Hand Wrung
- ProCell Wrung (Experimental): ProCell wrung refers to automated wringing surgical sponges by an FDA approved suction device (ProCell).
  Interventions: Device: ProCell Wrung

INTERVENTIONS:
Procedure: Hand Wrung — Hand wrung refers to manually wringing surgical sponges by hand.
  Arms: Hand Wrung
Device: ProCell Wrung — ProCell wrung refers to automated wringing surgical sponges by an FDA approved suction device (ProCell).
  Arms: ProCell Wrung

SUMMARY:
The purpose of this research study is to compare two methods of recovering blood from surgical sponges used during heart and lung surgeries. The two methods are: 1) manually wringing sponges by hand, and 2) automated wringing sponges by an FDA approved suction device. Both methods are already in use in heart and lung surgeries at University Hospitals at the discretion of the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing heart or lung transplant, redo sternotomy, aortic surgery, and/or multi-valve repairs/replacements; and
* At University Hospitals Cleveland Medical Center.

Exclusion Criteria:

* Patients with known bleeding disorders, including disseminated intravascular coagulation (DIC), prothrombin deficiency, factor V deficiency, factor VII deficiency, factor X deficiency, factor XI deficiency (hemophilia C), Glanzmann disease, hemophilia A, hemophilia B, idiopathic thrombocytopenic purpura (ITP), and Von Willebrand disease (types I, II, and III);
* Patients undergoing emergent or emergent salvage surgery; and
* Patients actively participating in another clinical trial which could affect outcomes.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Level of Plasma Free Hemoglobin | Baseline
  Level of plasma free hemoglobin will be measured at baseline.
Level of Plasma Free Hemoglobin | Post-Processing (Up to 120 Minutes)
  Level of plasma free hemoglobin will be measured post-processing.
Change in Volume of Blood | Baseline, Post-Processing (Up to 120 Minutes)
  Volume of blood will be measured at baseline and post-processing.

SECONDARY OUTCOMES:
Number of Fragmented Red Blood Cells | Baseline
  Number of fragmented red blood cells will be measured at baseline.
Number of Fragmented Red Blood Cells | Post-Processing (Up to 120 Minutes)
  Number of fragmented red blood cells will be measured post-processing.
Level of Lactate Dehydrogenase | Baseline
  Level of lactate dehydrogenase will be measured at baseline.
Level of Lactate Dehydrogenase | Post-Processing (Up to 120 Minutes)
  Level of lactate dehydrogenase will be measured post-processing.
Level of Haptoglobin | Baseline
  Level of haptoglobin will be measured at baseline.
Level of Haptoglobin | Post-Processing (Up to 120 Minutes)
  Level of haptoglobin will be measured post-processing.
Change in Weight of Surgical Sponge | Baseline, Post-Procedure (Up to 5 Minutes)
  Weight of surgical sponges will be measured at baseline and post-procedure.
Time to Wring Sponges | Up to 120 Minutes
  Time to wring sponges will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Arora, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No